CLINICAL TRIAL: NCT06527937
Title: A 2-Part, Phase 2, Open-Label, Randomized, Fixed Sequence Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Epinephrine After Single and Repeat Doses of DESF in Healthy Adults With Oral Allergy Syndrome (OASIS: Oral Anaphylm Symptom Intervention Study)
Brief Title: Pharmacokinetics Study of DESF in Adults With Oral Allergy Syndrome
Acronym: OASIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aquestive Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AQ109206
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2024-11

CONDITIONS: Allergic Reaction
MeSH Terms: conditions — Hypersensitivity | interventions — Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Doses of DESF and Intramuscular Manual Injection (Experimental): Single dose of DESF (12 mg) administered after allergen challenge (Treatment Period 1), followed by a single dose of intramuscular (IM) manual injection (0.3 mg) without allergen challenge after a 24-hour washout period (Treatment Period 2), followed by a single dose of DESF (12 mg) without allergen challenge after a 14-day washout period from Treatment Period 1.
  Interventions: Drug: DESF; Drug: Epinephrine Injection
- Repeat Doses of DESF and Intramuscular Manual Injection (Experimental): Repeat dose of DESF (24 mg [12 mg x 2]) administered after allergen challenge (Treatment Period 1), followed by a repeat dose of IM manual injection (0.6 mg [0.3 mg x 2]) without allergen challenge after a 24-hour washout period (Treatment Period 2), followed by a repeat dose of DESF (24 mg [12 mg x 2]) without allergen challenge after a 14-day washout period from Treatment Period 1.
  Interventions: Drug: DESF; Drug: Epinephrine Injection

INTERVENTIONS:
Drug: DESF — DESF administered in the sublingual space.
Drug: Epinephrine Injection — Epinephrine manual injection administered intramuscularly according to the approved prescribing information.

SUMMARY:
A 2-part open-label study to assess the pharmacokinetics (PK) and pharmacodynamics (PD) of epinephrine administered as single and repeat doses of DESF in healthy adults with oral allergy syndrome (OAS). In both parts, subjects undergo an oromucosal allergen challenge prior to administration of DESF according to randomization into two cohorts. In Part 1, there are three treatment periods evaluating single and repeat doses of study drug, DESF after an allergen challenge (Treatment Period 1), intramuscular (IM) injection without allergen challenge (Treatment Period 2), and DESF without allergen challenge (Treatment Period 3). In Part 2, there are two treatment periods evaluating single and repeat doses of study drug, DESF after an allergen challenge (Treatment Period 1) and intramuscular (IM) injection without allergen challenge (Treatment Period 2).

DETAILED DESCRIPTION:
This is a 2-Part, Phase 2, open-label, three-period, six-treatment, fixed sequence, stratified study conducted in healthy male and female adult subjects (age 18-55 years) who have oral allergy syndrome (OAS) designed to evaluate the pharmacokinetics (PK) of epinephrine administered as single and repeat doses of DESF with allergen-challenge induced oral physiological changes compared to the PK of epinephrine administered as single and repeat doses of intramuscular (IM) injection and single and repeat doses of DESF without allergen challenge. In both Part 1 and Part 2, all subjects undergo an allergen challenge prior to Treatment Period 1. Provided the allergen challenge elicits at least mild symptoms of oral physiological changes, subjects are randomized into one of two cohorts to receive either single or repeat doses of study drug throughout the study.

Allergen Challenge: The oromucosal allergen challenge begins approximately 20 minutes before the expected administration of DESF. Subjects have a single food allergen known to trigger an allergic reaction in the subject placed on their tongue for up to 15 minutes after initial exposure to upper and lower lips and gums. Subjects keep the allergen in place for up to 15 minutes until symptoms are reported. The subjects are monitored from the start of the allergen challenge to determine severity of symptoms. The allergen is then removed from the mouth and within 5 minutes subjects rate their symptoms and DESF is administered.

Part 1:

Up to 36 subjects will be enrolled in Part 1.

Treatment Period 1: Following the allergen challenge, subjects receive a single or repeat dose of DESF based on randomization.

Treatment Period 2: Subjects who complete Treatment Period 1 and a minimum 24-hour washout period receive either a single or repeat dose of manual IM epinephrine injection without an allergen challenge based on the randomization.

Treatment Period 3: Subjects who complete Treatment Period 1 and Treatment Period 2 undergo a minimum 14-day washout period from Treatment Period 1. Subjects are administered a single or repeat dose of DESF without an allergen challenge based on randomization.

Part 2:

Up to 12 subjects who have completed Part 1 (6 from each cohort) may continue to Part 2.

Treatment Period 1: Following the allergen challenge, subjects receive a single or repeat dose of DESF based on randomization in Part 1.

Treatment Period 2: Subjects who complete Treatment Period 1 and a minimum 24-hour washout period receive either a single or repeat dose of manual IM epinephrine injection without an allergen challenge based on the randomization.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent and capable of following the protocol-required guidelines.
* Healthy males and females 18 through 55 years of age.
* Body weight ≥50 kg for males and ≥45 kg for females.
* BMI ≥18 kg/m2 to ≤32 kg/m2.
* Known history of oral allergy syndrome in response to exposure to any of the allergens (e.g., apple, cherry, mango, melon, kiwi, celery, banana and/or carrot).
* Able to tolerate venipuncture.
* Subject has not had exposure to antihistamines within 3 days prior to the Screening visit.

Exclusion Criteria:

* Any current 'clinically significant' medical condition(s) that, in the opinion of the investigator, could confound the assessment of safety or impact assessments of PK and/or PD parameters or the safety of the subjects in the trial such as significant systemic neurological, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, oncologic and/or metabolic disease.
* Clinically significant laboratory results at Screening, including, but not limited to hemoglobin <11.5 g/dL for males or <10.5 g/dL for females.
* Clinically significant 12-lead ECG findings (at any time).
* Known history or presence of hypersensitivity or idiosyncratic reaction to DESF, epinephrine, or other drug substances with similar activity including intolerance or hypersensitivity to any component of DESF.
* Known history or presence of any disorder of the sublingual mucosa or any disease or condition which affects the normal production of saliva (e.g., xerostomia, Ehlers-Danlos syndrome, or Sjögren's syndrome) which, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results.
* Subject has a disorder of the sublingual mucosa that, in the opinion of the investigator, would impact or interfere with administration, retention or absorption of DESF.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 to 240 minutes post-dose
  Baseline Corrected Maximum Epinephrine Plasma Concentration occurring at Tmax (Time to reach maximum concentration)
AUC0-10 | 0 to 10 minutes
  Baseline Corrected Plasma Epinephrine Concentration-Time Curve from Time Zero to 10 minutes
AUC0-20 | 0 to 20 minutes
  Baseline Corrected Plasma Epinephrine Concentration-Time Curve from Time Zero to 20 minutes
AUC0-30 | 0 to 30 minutes
  Baseline Corrected Plasma Epinephrine Concentration-Time Curve from Time Zero to 30 minutes
AUC0-45 | 0 to 45 minutes
  Baseline Corrected Plasma Epinephrine Concentration-Time Curve from Time Zero to 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lee, MD, Principal Investigator — Frontage Clinical Services
Locations (1):
- Frontage Clinical Services, Inc., Secaucus, New Jersey, United States